CLINICAL TRIAL: NCT05730491
Title: Randomized Controlled Trial of an Internet-based Prevention Intervention for Parents With Irritable Bowel Syndrome
Brief Title: Online Social Learning Program for Parents With Irritable Bowel Syndrome: Raising Resilient Children
Acronym: REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R01HD107794-01 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome; Abdominal Pain
Keywords: social learning; cognitive behavioral therapy; prevention intervention; irritable bowel syndrome; solicitous behavior; protective factors; psychosocial intervention; abdominal pain; risk factors; illness behavior
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Illness Behavior | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either an attention educational control website or social learning cognitive behavioral therapy (SLCBT) prevention intervention. A control arm is necessary in order to evaluate the efficacy of the SLCBT intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are not informed of their condition assignment and both receive online programs focused on healthy child behaviors. Investigators are blinded & masked to study condition, and all outcomes are assessed via self-reported REDCap surveys. Care providers are not involved in the study (N/A).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Learning and Cognitive Behavioral Therapy (SLCBT) (Experimental)
  Interventions: Behavioral: Social Learning and Cognitive Behavioral Therapy (SLCBT)
- Attention Education Control (Placebo Comparator)
  Interventions: Behavioral: Attention Education Control

INTERVENTIONS:
Behavioral: Social Learning and Cognitive Behavioral Therapy (SLCBT) — Participants assigned to this group will complete an online program with 3 core skills, which will include strategies to promote wellness behaviors, use adaptive cognitive coping strategies, model wellness behaviors for their children, and determine when it is appropriate to take further action re: potential illness in their child. The website is interactive and self-guided. All participants will have access to the same resources and content, although based on responses to quizzes and skills practice questions, the automated feedback may differ slightly. The website includes treatment modules that share content via text, images, videos and recordings, a skills library that includes audio recordings of relaxation exercises, infographics to support skills practice, and behavioral assignments to record skills practice and receive automated feedback. Participants will review their knowledge at the end of each treatment module with brief quizzes.
  Arms: Social Learning and Cognitive Behavioral Therapy (SLCBT)
Behavioral: Attention Education Control — Participants assigned to the control group will receive access to a web program and complete 3 modules focused on child health and safety behaviors, such as sports and water safety. These participants will review written/visual content on the above topics, take quizzes to test knowledge gained, and will be provided with brief assignments to increase child safety behaviors. All participants assigned to the control group will have access to the same educational content.
  Arms: Attention Education Control

SUMMARY:
The goal of this clinical trial is to test efficacy of the REACH program in parents with irritable bowel syndrome (IBS) and their young children. The main question it aims to answer is:

-How can parents with IBS help their young kids develop healthy habits?

Participants will be asked to complete online surveys and to use a website. Researchers will compare results from parents who use one of two websites chosen by chance, like flipping a coin. One website focuses on child health and safety behaviors. The other website focuses on strategies to promote child wellness behaviors.

DETAILED DESCRIPTION:
To date, preventive interventions have not been applied to reduce intergenerational transmission of pain conditions. There are several reasons that abdominal pain presents an ideal model for this important work. Abdominal pain is the second most common recurrent pain complaint of childhood. It is associated with disruption of normal activity, including school attendance and poor quality of life, and is emotionally distressing for both children and parents. Research demonstrates that illness behaviors are linked to development of abdominal pain disorders in children.

The investigators hypothesize that a social learning intervention modified toward a preventive focus for parents with IBS who have young children, ages 4-7 years, will reduce risk factors (anxiety, catastrophizing, parenting stress) and increase protective factors (positive affect, social support), resulting in lower parental solicitous behaviors, fewer child abdominal pain symptoms, reduced child health care utilization, and better child physical, psychological, social, and school functioning. The objective of the current application is to test the efficacy of an early preventive intervention targeting parents with IBS whose young children are thus at higher risk for developing abdominal pain. To enhance potential for scalability and dissemination, and meet parental preferences, the intervention is delivered via the internet.

ELIGIBILITY:
Inclusion criteria for parents and their children (including biological/step-parents or legal guardians):

* Parent/caregiver at least 18 years old
* Parent diagnosed with IBS or idiopathic abdominal pain in the last five years OR
* Parent meets ROME criteria for IBS (abdominal pain at least weekly; pain related to defecation, change in stool frequency, and change in stool form at least 30% of the time)
* Is the parent primarily responsible for caring for the child on a day-to-day basis
* Child is 4 to 7 years old at the time of screening. If multiple children are present in the family, the parent will be asked to select one child for study participation.
* Child must currently live at least half of the time with the parent involved in intervention.
* Parent and child must reside in the U.S.

Exclusion criteria for parents and their children:

* Not able to read/speak/understand English.
* Child has a developmental disability that requires full-time special education
* Child has chronic abdominal pain (pain most/every day for more than 3 months)
* Child has a current doctor's diagnosis of a painful* gastrointestinal disorder like functional constipation, lactose/fructose/gluten intolerance, celiac disease, Inflammatory Bowel Disorder, etc. (*does not include nonpainful disorders like GERD)
* Child has another severe chronic disease such as juvenile arthritis, cancer, or other severe condition(s) requiring chronic medical treatment.
* Does not have regular access to the Internet on a desktop, tablet, phone, or laptop computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in parental encouragement of child illness behavior | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Assesses self-reported parental encouragement of child illness behavior. The Adult Responses to Child Symptoms (ARCS) has 29-items that load onto 3 subscales (Protectiveness, Monitoring/Encouragement, Minimization). Responses are rated on a 5-point scale ranging from "never" to "always." . Higher average scores indicate that the responses are more frequently used, and thus higher scores are less adaptive ways of responding.

SECONDARY OUTCOMES:
Change in anxiety | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent self-report. The Generalized Anxiety Disorder (GAD2) is one of the most frequently used diagnostic self-report scales for screening, diagnosis and severity assessment of anxiety disorders in adults. The scale is based on two items which are scored from 0 to 3, with higher scores indicating greater anxiety symptoms.
Change in pain catastrophizing | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent self-report. Pain Catastrophizing Scale, is a 13-item measure that assesses catastrophizing thoughts or feelings accompanying the experience of pain. Respondents are asked to reflect on past painful experiences and to indicate the degree to which each of the 13 thoughts or feelings were experienced when in pain. Responses are from 0 (not at all) to 4 (all the time) with higher scores indicating higher levels of catastrophizing.
Change in positive and negative affect | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent self-report. Positive and Negative Affect Schedule (PANAS) is a widely used self-report measure that is made up of two mood scales. One 10-item scale measures positive affect and the other 10-item scale measures negative affect on a 5-point Likert scale. Scores range from 10-50 for each scale with higher scores indicating high levels of positive or negative affect.
Change in perceived social support | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent self-report. Perceived Social Support will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS). This scale consists of 12 items that measure the extent of social support received from 3 sources: friends, family, and significant others. Types of social support assessed by the MSPSS include emotional, tangible, informational, social network support, and esteem. Scores range from 12 to 84 with higher scores indicating greater social support.
Change in health-related quality of life | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent proxy report and child self-report (ages 7+). The Pediatric Quality of Life Inventory (PedsQL) is a brief measure of health-related quality of life in children. The measure can be completed by parents (the Proxy Report) for children as young as age 2 years. The 23 items in the PedsQL comprise four Generic Core Scales: Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items), and School Functioning (5 items). Two Summary Scores can be computed (the Psychosocial Health Summary Score and the Physical Health Summary Score), as well as a Total Scale Score. Scores range from 0-100, with higher scores indicating better quality of life.
Change in health care costs | Baseline, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parents will complete the Client Service Receipt Inventory (CSRI), a validated comprehensive inventory of health care services incurred due to the child's symptoms that uses a standard response timeframe of the past 6 months. In the CSRI, parents report on three sources of health care costs: direct medical service use, direct non-medical costs, and indirect costs. In order to better estimate costs, monetary values will be assigned to health resources use and productivity time loss data captured in the CSRI. All expenditures will be converted to 2023 dollars using the medical care component of the Consumer Price Index available from the Bureau of Labor Statistics. Costs will be aggregated across the three sources to derive total costs for analyses.
Change in pain intensity | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent proxy report and child self-report (ages 7+). The Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity form includes three items assessing child's pain intensity in the past 7 days.
Change in somatic symptoms | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent proxy report. The Children's Somatic Symptoms Inventory (CSSI-8) includes 8 items assessing the severity of a child's nonspecific somatic symptoms. The set of GI symptoms (pain, nausea, upset stomach) are used to measure GI symptom severity.
Change in abdominal pain symptoms | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent proxy report. The ROME Functional Abdominal Pain questions include 5 items assessing ROME criteria for upper and lower functional abdominal pain - frequency, severity, location, and association with eating (lower only).
Change in depressive symptoms | Baseline, 4-6 weeks, 6 months post-intervention, 12 months post-intervention, and 18 months post-intervention
  Parent self-report. The Patient Health Questionnaire (PHQ2) includes 2 items inquiring about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks.
Change in parenting stress | Baseline
  Parent self-report. The Daily Parenting Hassles Scale is a 20-item scale that assesses parent burden in meeting the needs of their children and troublesome behavior of children. Subscales include challenging behavior and parenting tasks.
Number of treatment contacts | 0-6 weeks
  The administrative backend of the intervention programs has a tracking system for recording use of the program. Specifically, we will measure: 1) logins to the program, 2) completed treatment modules, and 3) completed assignments.
Treatment acceptability | 4-6 weeks
  The TEI-SF is a 9-item measure that assesses treatment acceptability and satisfaction. Select items were adapted to be specific to a parenting prevention program (e.g., "I find this intervention to be an acceptable way of dealing with young children's health"). Items are rated on a 5-point scale (1 = 'strongly disagree', 5 = 'strongly agree') and summed to create a total score, with higher scores indicating higher acceptability and satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy RL, Murphy TB, van Tilburg MAL, Kuklinski MR, Bailey JA, Aalfs H, Badillo I, Diakhate H, Palermo TM. Protocol for a randomized controlled trial of an internet-based prevention intervention for young children at-risk for functional abdominal pain. Trials. 2024 Aug 19;25(1):549. doi: 10.1186/s13063-024-08371-8. PMID 39160566